CLINICAL TRIAL: NCT00000796
Title: A Prospective Study of Multidrug Resistance and a Pilot Study of the Safety of and Clinical and Microbiologic Response to Levofloxacin in Combination With Other Antimycobacterial Drugs for Treatment of Multidrug-Resistant Pulmonary Tuberculosis (MDRTB) in HIV-Infected Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 238; CPCRA 026; 11215 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Tuberculosis
Keywords: Isoniazid; Tuberculosis, Pulmonary; Pyrazinamide; Pyridoxine; Ofloxacin; Rifampin; AIDS-Related Opportunistic Infections; Drug Therapy, Combination; Ethambutol; Clofazimine; Acquired Immunodeficiency Syndrome; Amikacin; Drug Resistance, Microbial; Cycloserine; Capreomycin Sulfate; Ethionamide; Aminosalicylic Acids; Streptomycin; p-Aminosalicylic Acid
MeSH Terms: conditions — HIV Infections; Tuberculosis; Tuberculosis, Pulmonary; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome | interventions — Cycloserine; Ethionamide; Capreomycin; Aminosalicylic Acid; Streptomycin; Ethambutol; Amikacin; Isoniazid; Pyrazinamide; Pyridoxine; Levofloxacin; Rifampin; Clofazimine

INTERVENTIONS:
Drug: Cycloserine
Drug: Ethionamide
Drug: Capreomycin sulfate
Drug: Aminosalicylic acid
Drug: Streptomycin sulfate
Drug: Ethambutol hydrochloride
Drug: Amikacin sulfate
Drug: Isoniazid
Drug: Pyrazinamide
Drug: Pyridoxine hydrochloride
Drug: Levofloxacin
Drug: Rifampin
Drug: Clofazimine

SUMMARY:
To determine the demographic, behavioral, clinical, and geographic risk factors associated with the occurrence of multidrug-resistant pulmonary tuberculosis (MDRTB). To evaluate the clinical and microbiological responses and overall survival of MDRTB patients who are treated with levofloxacin-containing multiple-drug regimens chosen from a hierarchical list. Per 9/28/94 amendment, to assess whether persistent or recurrent positive sputum cultures of patients who show failure or relapse are due to the same strain or reinfection with a new strain.

Among TB patients, there has been an increase in progressive disease due to the emergence of antimycobacterial drug-resistant strains of Mycobacterium tuberculosis. Failure to identify patients at high risk for MDRTB increases the hazard for both treatment failure and development of resistance to additional therapeutic agents. Efforts to improve survival in patients with MDRTB will depend on improved methods of assessing the risk of acquisition of MDRTB and identifying drug susceptibility patterns in a timely fashion.

DETAILED DESCRIPTION:
Among TB patients, there has been an increase in progressive disease due to the emergence of antimycobacterial drug-resistant strains of Mycobacterium tuberculosis. Failure to identify patients at high risk for MDRTB increases the hazard for both treatment failure and development of resistance to additional therapeutic agents. Efforts to improve survival in patients with MDRTB will depend on improved methods of assessing the risk of acquisition of MDRTB and identifying drug susceptibility patterns in a timely fashion.

Patients are asked a series of questions to determine epidemiologic factors that may be predictive of MDRTB. Patients who are determined to be at low risk for MDRTB will be referred to another TB treatment protocol (ACTG 222), if appropriate. Patients suspected of having primary or acquired MDRTB or those with confirmed MDRTB will be offered a regimen of anti-TB therapy from a hierarchically ordered list of drugs, based on the patient's resistance status (suspect primary MDRTB, suspect acquired MDRTB, or confirmed MDRTB). The hierarchical list is as follows: isoniazid, rifampin, ethambutol, streptomycin, levofloxacin, ethionamide, cycloserine, capreomycin, aminosalicylic acid, and clofazimine. Treatment will be administered daily for at least 6 months, then on an intermittent schedule at the clinician's discretion. Patients with confirmed MDRTB (defined as known resistance to at least isoniazid and rifampin within 6 months prior to study entry) will receive a minimum of 18 months of treatment following sputum culture conversion. Follow-up is performed every 4 weeks for 8 weeks, and then every 8 weeks.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Working diagnosis of HIV infection.
* Working diagnosis of pulmonary TB.

Per 08/02/94 amendment, patients with confirmed MDRTB or known susceptibilities for the current episode at baseline are not eligible for the epidemiologic study only.

FOR TREATMENT PILOT:

* Positive sputum AFB smear (or a positive sputum culture for TB within 6 months prior to study entry).
* Assessment of suspect primary, suspect acquired, AND/OR confirmed MDRTB.
* Life expectancy of at least 2 weeks.
* Age >= 18 years for suspect MDRTB. Age >= 13 years for confirmed MDRTB.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Known hypersensitivity or resistance to quinolones.
* Other disorders or conditions for which the study drugs are contraindicated.

Prior Medication:

Excluded:

* More than 6 weeks total therapy within 3 months prior to study entry using three or more drugs effective against the isolates. (Per 08/02/94 amendment, patients from protocol ACTG 222/CPCRA 019 who have MDRTB are eligible for rollover to this study regardless of treatment duration on ACTG 222/CPCRA 019.)

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 525
Dates: Study Completion 1998-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Telzak E, Study Chair; Benson C, Study Chair; Chirgwin K, Study Chair; Sepkowitz K, Study Chair
Locations (21):
- United States (21):
  - Cook County Hosp, Chicago, Illinois
  - Henry Ford Hosp, Detroit, Michigan
  - Interfaith Med Ctr, Brooklyn, New York
  - SUNY / Health Sciences Ctr at Brooklyn, Brooklyn, New York
  - Beth Israel Med Ctr, New York, New York
  - Clinical Directors Network of Region II, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Saint Clare's Hosp and Health Ctr, New York, New York
  - Cornell Univ Med Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Columbia Presbyterian Med Ctr, New York, New York
  - Harlem AIDS Treatment Group / Harlem Hosp Ctr, New York, New York
  - Bronx Lebanon Hosp Ctr, The Bronx, New York
  - Bronx Municipal Hosp Ctr/Jacobi Med Ctr, The Bronx, New York
  - Comprehensive Health Care Ctr / Bronx Municipal Hosp, The Bronx, New York
  - Montefiore Drug Treatment Ctr / Bronx Municipal Hosp, The Bronx, New York
  - Montefiore Family Health Ctr / Bronx Municipal Hosp, The Bronx, New York
  - Samaritan Village Inc / Bronx Municipal Hosp, The Bronx, New York
  - Jack Weiler Hosp / Bronx Municipal Hosp, The Bronx, New York
  - Montefiore Med Ctr / Bronx Municipal Hosp, The Bronx, New York
  - North Central Bronx Hosp / Bronx Municipal Hosp, The Bronx, New York

REFERENCES:
- [Background] Telzak EE, Chirgwin K, Nelson E, Matts J, Benson C, Sepkowitz K, Perlman D, El-Sadr W. Predictors for multidrug-resistant tuberculosis (MDRTB) among HIV-infected patients and response to specific MDRTB drug regimens. Conf Retroviruses Opportunistic Infect. 1997 Jan 22-26;4th:184 (abstract no 647)
- [Background] Telzak EE, Chirgwin KD, Nelson ET, Matts JP, Sepkowitz KA, Benson CA, Perlman DC, El-Sadr WM. Predictors for multidrug-resistant tuberculosis among HIV-infected patients and response to specific drug regimens. Terry Beirn Community Programs for Clinical Research on AIDS (CPCRA) and the AIDS Clinical Trials Group (ACTG), National Institutes for Health. Int J Tuberc Lung Dis. 1999 Apr;3(4):337-43. PMID 10206505